CLINICAL TRIAL: NCT05756842
Title: The Effect of a Honey-based Gel Supplement From the Wider Area of Pindos on Human Health and Oxidative Stress Biomarkers
Brief Title: Honey Consumption, Oxidative Stress and Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Z. Jamurtas, Professor, University of Thessaly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UTH-HoneyGel
Record Dates: First submitted 2023-02-18; First posted 2023-03-06 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Oxidative Stress
Keywords: Oxidative stress; Honey; Antioxidants; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Honey-based gel consumption (Experimental): A honey-based gel will be administered to participants in this arm.
  Interventions: Dietary Supplement: Honey-based gel supplementation

INTERVENTIONS:
Dietary Supplement: Honey-based gel supplementation — 70 g/day of a honey-based gel divided into 2 equal doses of 35 gr (in the morning and evening) for a total duration of 14 days

SUMMARY:
The aim of the present clinical study is to estimate the efficacy of a honey-based gel, derived from the wider area of Pindos in Greece, in regulating oxidative stress biomarkers and the physiological profile of healthy adults.

DETAILED DESCRIPTION:
Introduction: Honey contains about 200 compounds such as sugars, proteins, vitamins, water, free amino acids, enzymes, minerals, and many phytochemicals. Due to its composition, enriched with many bioactive ingredients, several studies have established its antimicrobial, antiviral, anticancer, antidiabetic and antioxidant properties. This multilayer activity of honey has been proposed for the protection against pathologies interrelated with the cardiovascular, nervous, respiratory, and gastrointestinal system.

Purpose: This study aims to investigate the effects of a novel natural honey-based gel consumption on oxidative stress biomarkers, blood chemistry and physiological characteristics in healthy individuals.

Methodology: A total of 20 healthy men and women will participate in the study. Participants will give their informed consent after they will be informed about the purposes, procedures, risks and benefits associated with the study. Participants will consume 70 g/day of the honey-based gel, distributed in 2 equal doses (in the morning and evening) for 14 days. At baseline and post-intervention, volunteers will be assessed for their physiological profile and will provide a resting blood sample for the assessment of oxidative stress and blood chemistry biomarkers as well as their physiological profile. Participants will be asked to record their diet for 3 days prior to the study and they will be asked to follow the same dietary pattern for 3 days before the post-intervention assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Individuals aged 18-65 years
* Non-smokers

Exclusion Criteria:

* Musculoskeletal injury
* Dietary supplements
* Medication
* Allergy in bee pollen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in glutathione concentration of erythrocytes | Change from baseline to 14 days
  Glutathione concentration will be analyzed in erythrocytes by spectrophotometry
Change in catalase enzyme activity of erythrocytes | Change from baseline to 14 days
  Catalase enzyme activity will be analyzed in erythrocytes by spectrophotometry
Change in total antioxidant capacity of plasma | Change from baseline to 14 days
  Total antioxidant capacity will be analyzed in plasma by spectrophotometry
Change in thiobarbituric acid reactive substances of plasma | Change from baseline to 14 days
  Thiobarbituric acid reactive substances will be analyzed in plasma by spectrophotometry
Change in protein carbonyls of plasma | Change from baseline to 14 days
  Protein Carbonyls will be analyzed in plasma by spectrophotometry
Change in body weight | Change from baseline to 14 days
  Body weight will be measured using a digital scale
Change in body fat | Change from baseline to 14 days
  Body fat will be measured by bioelectrical impedance analysis
Change in resting heart rate | Change from baseline to 14 days
  Resting heart rate will be measured using a heart rate sensor
Change in diastolic and systolic blood pressure | Change from baseline to 14 days
  Diastolic and systolic blood pressure will be measured using a manual sphygmomanometer
Change in waist and hip circumference | Change from baseline to 14 days
  Waist and hip circumference will be assessed using a tape measure
Change in complete blood count | Change from baseline to 14 days
  White blood cells, lymphocytes, monocytes, granulocytes, red blood cells and platelets will be analyzed in whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Z. Jamurtas, Professor, Study Director — University of Thessaly
Locations (1):
- Exercise Biochemistry, Physiology and Nutrition Laboratory, Department of Physical Education and Sport Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohd Kamal DA, Ibrahim SF, Kamal H, Kashim MIAM, Mokhtar MH. Physicochemical and Medicinal Properties of Tualang, Gelam and Kelulut Honeys: A Comprehensive Review. Nutrients. 2021 Jan 10;13(1):197. doi: 10.3390/nu13010197. PMID 33435215
- [Background] Escuredo O, Miguez M, Fernandez-Gonzalez M, Carmen Seijo M. Nutritional value and antioxidant activity of honeys produced in a European Atlantic area. Food Chem. 2013 Jun 1;138(2-3):851-6. doi: 10.1016/j.foodchem.2012.11.015. Epub 2012 Nov 17. PMID 23411187
- [Background] Schramm DD, Karim M, Schrader HR, Holt RR, Cardetti M, Keen CL. Honey with high levels of antioxidants can provide protection to healthy human subjects. J Agric Food Chem. 2003 Mar 12;51(6):1732-5. doi: 10.1021/jf025928k. PMID 12617614